CLINICAL TRIAL: NCT00218608
Title: Disulfiram for Cocaine Abuse in Methadone- Patients
Brief Title: Disulfiram for Treating Cocaine Dependence in Individuals Maintained on Methadone
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIDA-13441-1; R01-13441-1; DPMC
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2012-01

CONDITIONS: Cocaine-Related Disorders; Opioid-Related Disorders
Keywords: Cocaine Abuse
MeSH Terms: conditions — Cocaine-Related Disorders; Opioid-Related Disorders | interventions — Disulfiram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator): Placebo (microcrystalline cellulose) was suspended in the methadone during weeks 3-14.
  Interventions: Drug: Disulfiram
- Disulfiram at 62.5 mg (Active Comparator): Disulfiram at 62.5 mg was suspended in the methadone during weeks 3-14.
  Interventions: Drug: Disulfiram
- Disulfiram at 125 mg (Active Comparator): Disulfiram at 125 mg/day was suspended in methadone during weeks 3-14.
  Interventions: Drug: Disulfiram
- Disulfiram at 250 mg (Active Comparator): Disulfiram at 250 mg/day was suspended in methadone during weeks 3-14.
  Interventions: Drug: Disulfiram

INTERVENTIONS:
Drug: Disulfiram — Disulfiram at 0, 62.5, 125 and 250 mg/day were administered during weeks 3-14
  Other Names: Antabuse

SUMMARY:
Cocaine is an extremely addictive stimulant drug that directly affects the brain. It is used in several different forms and can be snorted, smoked, or injected to achieve the desired effect. Cocaine users are at risk for many health problems, both directly and indirectly related to the effects of cocaine. Disulfiram, a drug used to treat chronic alcoholism, may be effective in reducing cocaine use. This study will evaluate the effectiveness of three different doses of disulfiram in treating cocaine dependence in opioid- and cocaine-dependent individuals maintained on methadone.

DETAILED DESCRIPTION:
Despite the harm that cocaine can cause to the body, its abuse is widespread. It is the cause of more visits to hospital emergency rooms nationwide than any other illegal drug. Effective treatments for cocaine and opiate addictions are essential to the decline of cocaine- and opiate-related disorders. Unfortunately, cocaine use remains prevalent among participants in many opioid maintenance programs. The addition of other medications to methadone maintenance may prove helpful in reducing cocaine use. Disulfiram, a drug used to treat chronic alcoholism, causes unpleasant effects when even small amounts of alcohol are consumed. This study will evaluate the effectiveness of three different doses of disulfiram in treating cocaine dependence in opioid- and cocaine-dependent individuals maintained on methadone.

Participants in this double blind study will be randomly assigned to receive either disulfiram at one of three dosage levels (62.5, 125, 250 mg/day) or placebo for 14 weeks. During the first 2 weeks, doses of methadone plus either disulfiram or placebo will be administered until the assigned maintenance dose is achieved. This dosage level will be maintained for the duration of the study. Participants will be required to report to the study site Monday through Saturday of each week for assessments and to receive medication. They will receive a take-home dose of medication for Sunday. In addition, participants will receive a weekly session of cognitive-behavioral therapy. Urine samples will be collected three times a week to assess drug use. At the end of the study, participants will undergo a 4- to 6-week detoxification period in which they will gradually discontinue the use of methadone and disulfiram. All participants have the option to request transfer to a local methadone maintenance program instead of undergoing detoxification.

Enrollment has been completed and no subjects are active. Data analyses are being conducted at this time.

ELIGIBILITY:
Inclusion Criteria:

* History of cocaine use at least once a week during the month prior to study entry
* Urine screen tests positive for cocaine
* Meets DSM-IV criteria for opioid- and cocaine-dependence
* Urine toxicology screen tests negative for benzodiazepines prior to beginning methadone treatment

Exclusion Criteria:

* Current drug or alcohol dependence other than opiates, cocaine, or tobacco
* Significant medical condition, such as abnormal liver function (with laboratory findings greater than three times normal), active hepatitis, or high blood pressure
* Current cardiac condition
* Occult coronary artery disease
* At high risk for cardiovascular disease, seizure disorders, or any other significant underlying medical condition that may make treatment with disulfiram or methadone unsafe
* Meets DSM-IV psychiatric diagnostic criteria for lifetime schizophrenia, bipolar disorder, or other psychotic disorders
* Currently suicidal or homicidal
* Currently taking a prescribed psychotropic medication that cannot be discontinued
* Pregnant
* Currently taking metronidazole or clotrimazole

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2001-04; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Cocaine use | 14 wks
  Urine toxicology screens were conducted thrice-weekly for 14 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Alison Oliveto, PhD, Principal Investigator — UAMS
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States